CLINICAL TRIAL: NCT03344341
Title: A 24-Week, Multicenter, Randomized, Parallel-group, Open-label, Active Controlled Phase IV Study to Assess the Efficacy and Safety of Dapagliflozin as Monotherapy Compared With Acarbose in Drug-Naive Patients With Type 2 Diabetes Mellitus (T2DM) in China
Brief Title: A Phase IV Study in Drug-Naive Patients With T2DM in China
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study overall progress behind of scheduled timeline. Study was terminated early due to company decision.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1690C00060
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Acarbose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin is started from 5 mg once a day, taken orally in the morning, before or after breakfast. From the third week, the dose will be increased to 10 mg once a day and last to the end of the study.
  Interventions: Drug: Dapagliflozin
- Acarbose (Active Comparator): Acarbose is started from 50 mg once a day at dinner during the first week, titrated up to 50 mg twice a day at lunch and dinner in the second week, 50 mg three times a day at three meals in the third week, and 100 mg three times a day till the end of the study.
  Interventions: Drug: Acarbose

INTERVENTIONS:
Drug: Dapagliflozin — Starting dose of dapagliflozin is 5 mg once daily, taken orally in the morning, before or after breakfast. From the third week,the dose can be increased to 10 mg once daily, and last to the end of the study.
  Arms: Dapagliflozin
Drug: Acarbose — Acarbose was started from 50 mg once a day at dinner during the first week and titrated up to 50 mg twice a day at lunch and dinner in the second week, 50 mg three times a day at three meals in the third week, and 100 mg three times a day till the end of the study.
  Arms: Acarbose

SUMMARY:
This is a 24-week, multicenter, randomized, open-label, parallel-group, active controlled Phase IV study to assess the efficacy and safety of Dapagliflozin as monotherapy compared with Acarbose in patients with T2DM who were inadequately controlled with diet and exercise.

The study is designed to evaluate the efficacy and safety of dapagliflozin monotherapy compared with acarbose monotherapy in patients with T2DM inadequately controlled with diet and exercise.

DETAILED DESCRIPTION:
1. Study design This is a 24-week, multicenter, randomized, open-label, parallel-group, active controlled Phase IV study The open-label study design rather than double-blind is considered due to the difficulty of placebo supply. The primary efficacy endpoint will be blinded to both patients and investigators, so the measurements as well as the management of the patients will not be impacted by the design of open-label.

The study is powered to show non-inferiority of dapagliflozin versus acarbose regarding with HbA1c reduction.

A non-inferiority margin of 0.25% for the difference of the reduction in HbA1c is considered in the study.

1. Primary and secondary outcome variables In the clinical guidelines for type 2 diabetes, HbA1c is recommended as gold standard for determination of glycemic control and is therefore chosen as the primary outcome variable. Certain secondary outcome variables have been selected for additional assessment because of their clinical relevance and importance.
2. Dosing and study duration Dapagliflozin will be started from 5 mg once a day, taken orally in the morning, before or after food. In patients tolerating dapagliflozin 5 mg once a day, the dose will be increased to 10 mg once a day from the second week.

Acarbose will be started from 50 mg once a day at dinner during the first week and titrated up to 50 mg twice a day at lunch and dinner in the second week, 50 mg three times a day at three meals in the third week, and 100 mg three times a day from the fourth week onwards.

The dosing in study is in line with the local labels for dapagliflozin and acarbose.

Treatment duration of 24 weeks is considered to be adequate to establish glycemic efficacy of dapagliflozin monotherapy compared with acarbose monotherapy in lowering blood glucose indicated by HbA1c change in patients with T2DM inadequately controlled with diet and exercise.

2. Benefit/risk and ethical assessment According to the available data so far, glucose lowering effect of dapagliflozin is associated with a favourable safety and tolerability profile, and accompanied with a slightly increased risk of genital infection and urinary tract infection [9, 10].

Acarbose is the most widely used oral anti-diabetic drug in china. The common side effects of acarbose treatment are flatulence, borborygmus and diarrhoea, according to the prescribing information and clinical experience from physicians.

The treatment regimens in the study are in line the prescribing information for dapagliflozin and acarbose. Patients with potential contraindications or not considered to get benefit from dapagliflozin or acarbose treatment will be excluded from the study by the inclusion/exclusion criteria set in the study. And the patient safety will be closely monitored in the study by Adverse events/Serious Adverse events collecting and assessment, laboratory testing, ECG, glucometer, vital sign and physical examination.

Overall, the study drugs investigated and the study design is considered to have a favorable benefit-risk profile in the treatment of patients with T2DM.

Methods for assigning treatment groups A block stratified randomization method will be used to assign patients to the treatment groups in this study. Patients will be randomized 1:1 to treatment groups via a central randomization system (interactive voice / web response system [Interactive Voice Response System/Interactive Web Response System])(IVRS/IWRS), and drug will be dispensed accordingly.

The study population will be stratified based on the level of HbA1c at baseline (HbA1c < 8.0%、≥ 8.0% ~ < 9.0% and ≥9.0%)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed within the past 12 months with T2DM according to 1999 World Health Organization(WHO) criteria.
2. Men and women aged at least 18 years at screening.
3. Either not received oral anti-diabetic drugs or had been on short-term (1 month) treatment that had been discontinued 3 months before enrolment.
4. HbA1c ≥ 7.5% and ≤ 10.5% at screening and HbA1c ≥ 7.0% and ≤ 10.5% at pre-randomization visit.
5. FPG ≤ 13.3 mmol/L (≤ 240 mg/dL) .
6. BMI≥18.5 kg/m2 and ≤ 45.0 kg/m2 .
7. C-peptide ≥0.33nmol/L(≥1.0 ng/mL).
8. Able and willing to provide written informed consent and to comply with the study.

Exclusion Criteria:

1. Women who are pregnant, intending to become pregnant during the study period, currently lactating females, or women of child-bearing potential not using highly effective, medically approved birth control methods.
2. Diagnosis or history of:

   a. Acute metabolic diabetic complications such as ketoacidosis or hyperglycemic hyperosmolar state b. Diabetes insipidus.
3. Requirement for insulin therapy. Symptoms of poorly controlled diabetes, including but not limited to, marked polyuria and polydipsia with >10% weight loss during the 3 months before enrollment.
4. Triglycerides (fasting) > 9.3 mmol/L (> 800 mg/dL).
5. Patients with clinically apparent hepatobiliary disease, including but not limited to chronic active hepatitis and/or severe hepatic insufficiency. Alanine Aminotransferase(ALT) or Aspartate Aminotransferase(AST) > 3x upper limit of normal (ULN), or serum total bilirubin (TB) >34.2 μmol/L (>2 mg/dL).
6. Patients with following renal disease history or renal disease related features:

   1. History of unstable or rapidly progressing renal disease;
   2. Patients with moderate /severe renal impairment or end-stage renal disease (eGFR< 60 mL/min/1.73 m2);
   3. Urinary albumin: creatinine ratio >1800 mg/g;
   4. Serum creatinine (Cr) ≥133 μmol/L (≥1.50 mg/dL) for male subjects; Serum Cr≥124 μmol/L (≥1.40 mg/dL) for female subjects;
   5. Conditions of congenital renal glycosuria.
7. Severe uncontrolled hypertension defined as SBP ≥180 mmHg and/or BP ≥110 mmHg; Patients with SBP < 95mmHg.
8. Any of the following cardiovascular diseases within 6 months of the enrollment visit:

   1. Myocardial infarction;
   2. Cardiac surgery or revascularization (coronary artery bypass graft/percutaneous transluminal coronary angioplasty);
   3. Unstable angina;
   4. Congestive heart failure New York Heart Association Class III or IV;
   5. Transient ischemic attack or significant cerebrovascular disease.
9. History of gastrointestinal disease or surgery including Roemheld Syndrome, severe hernia, intestinal obstruction, intestinal ulcer, gastroenterostomy, enterectomy, bariatric surgery or lap-band procedure.
10. Malignancy within 5 years of the enrollment visit (with the exception of treated basal cell or treated squamous cell carcinoma).
11. Known immunocompromised status, including but not limited to, individuals who had undergone organ transplantation or acquired immunodeficiency syndrome (AIDS).
12. Any subject who, in the judgment of the investigator, was at risk for dehydration or volume depletion that might affect the interpretation of efficacy or safety data.
13. History of bone fracture secondary to diagnosed severe osteoporosis.
14. Currently unstable or serious cardiovascular, renal, hepatic, hematologic, oncologic, endocrine, psychiatric, or rheumatic diseases as judged by the Investigator.
15. Replacement or chronic systemic corticosteroid therapy, defined as any dose of systemic corticosteroid taken for >4 weeks within 3 months before enrollment visit.
16. Administration of sibutramine, phentermine, orlistat, rimonabant, benzphetamine, diethylpropion, methamphetamine, or phendimetrazine within 30 days of enrollment visit.
17. Any subject who was currently abusing alcohol or other drugs or had done so within the last 6 months.
18. Donation of blood or blood products, blood transfusion, or participation in a clinical study requiring withdrawal of >400 mL of blood during the 6 weeks before the enrollment visit.
19. History of hypersensitivity reaction to dapagliflozin or acarbose. Allergies or contraindication to the contents of dapagliflozin tablets or acarbose tablets.
20. Previous participation in a clinical trial with dapagliflozin.
21. Administration of any other investigational drug within 30 days of planned enrollment to this study, or within 5 half-life periods of other investigational drugs.
22. Subject is, in the judgment of the Investigator, unlikely to comply with the protocol or has any severe concurrent medical or psychological condition that may affect the interpretation of efficacy or safety data.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbA1c at Week 24 | At week 24
  Which will be derived using the HbA1c (%) at week 24 minus HbA1c (%) at baseline.

SECONDARY OUTCOMES:
Percentage of patients at Week 24 with reduction of HbA1c≥0.5%, body weight≥3% and SBP ≥3mmHg from baseline | From baseline to week 24
  Which will be derived using the number of patients who have reduction in HbA1c ≥ 5%, and body weight ≥3% and SBP ≥3 mmHg compared to baseline divided by the total number of patients.
Percentage of patients achieving HbA1c<7.0% | From baseline to week 24
  Which will be derived using the number of patient who have the HbA1c (%) < 7.0% after 24 weeks treatment divided by the total number of patients.
Percentage of patients with reduction of HbA1c≥0.5% | From baseline to week 24
  Which will be derived using the number of patients who have reduction in HbA1c≥0.5% after 24 weeks compared to baseline divided by the total number of patients.
Absolute change from baseline in fasting plasma glucose (FPG) | From baseline to week 24
  Which will be derived using the value of fasting plasma glucose (FPG) at post-baseline visits minus the value at baseline
Absolute change from baseline in 2h postprandial glucose (PPG) | From baseline to week 24
  Which will be derived using the value of 2h postprandial glucose (PPG) at the post-baseline visits minus the value at baseline
Absolute change from baseline in body weight | From baseline to week 24
  Which will be derived using the value of the body weight at the post-baseline visits minus the value at baseline
Percentage of patients with reduction of body weight ≥3% | From baseline to week 24
  Which will be derived using the number of patients who have reduction in body weight≥3% after 24 weeks compared to baseline divided by the total number of patients.
Absolute change from baseline in systolic blood pressure (SBP) | From baseline to week 24
  Which will be derived using the value of the systolic blood pressure at the post-baseline visits minus the value at baseline
Percentage of patients with reduction of SBP ≥3 mmHg | From baseline to week 24
  Which will be derived using the number of patients who have reduction in SBP ≥3 mmHg after 24 weeks compared to baseline divided by the total number of patients.

OTHER OUTCOMES:
Homeostasis model assessment-β | From baseline to week 24
  Which will be used to evaluate the beta cell function.
HOMA-IR | From baseline to week 24
  Which will be used to evaluate the insulin sensitivity
The difference of the number between tablets taken and tablets prescribed | From baseline to week 24
  Which will be derived using the number of tablets dispensed minus the number of tablets returned

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, Study Chair — Shanghai 6th People's Hospital
Locations (16):
- China (16):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Tianjin
  - Research Site, Xi'an
  - Research Site, Yinchuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Cefalu, W.T., et al., Dapagliflozin's Effects on Glycemia and Cardiovascular Risk Factors in High-Risk Patients With Type 2 Diabetes: A 24-Week, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study With a 28-Week Extension. Diabetes Care, 2015. 38(7): p. 1218-27. 2. Yang, W., et al., Prevalence of diabetes among men and women in China. N Engl J Med, 2010. 362(12): p. 1090-101. 3. Ji, L., et al., Primacy of the 3B approach to control risk factors for cardiovascular disease in type 2 diabetes patients. Am J Med, 2013. 126(10): p. 925.e11-22. 4. 中华医学会糖尿病学分会, 中国2型糖尿病防治指南(2013年版). 中华糖尿病杂志, 2014. 06((07): p. 447-498. 5. Komoroski, B., et al., Dapagliflozin, a novel, selective SGLT2 inhibitor, improved glycemic control over 2 weeks in patients with type 2 diabetes mellitus. Clin Pharmacol Ther, 2009. 85(5): p. 513-9. 6. Henry, R.R., et al., Dapagliflozin, metformin XR, or both: initial pharmacotherapy for type 2 diabetes, a randomised controlled trial. Int J Clin Pract, 2012. 66(5): p. 446-56. 7. Nauck, M.A., et al., Dapagliflozin versus glipizide as add-on therapy in patients with type 2 diabetes who have inadequate glycemic control with metformin: a randomized, 52-week, double-blind, active-controlled noninferiority trial. Diabetes Care, 2011. 34(9): p. 2015-22. 8. 中华医学会糖尿病分会, 中国2型糖尿病防治指南2013年版. 9. Johnsson, K.M., et al., Urinary tract infections in patients with diabetes treated with dapagliflozin. J Diabetes Complications, 2013. 27(5): p. 473-8. 10. Johnsson, K.M., et al., Vulvovaginitis and balanitis in patients with diabetes treated with dapagliflozin. J Diabetes Complications, 2013. 27(5): p. 479-84.